CLINICAL TRIAL: NCT04996693
Title: On Dose Efficiency of Modern CT-scanners in Chest Scans- a Prospective, Randomized Study
Brief Title: On Dose Efficiency of Modern CT-scanners in Chest Scans
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Augsburg (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 21-0368
Record Dates: First submitted 2021-07-23; First posted 2021-08-09 (Actual); Last update posted 2023-11-22 (Actual); Status verified 2023-11

CONDITIONS: Pneumonia; Lung Cancer; Pulmonary Embolism; Pulmonary Disease; Aortic Stenosis
Keywords: Spectral CT; Computed Tomography; Dose efficiency
MeSH Terms: conditions — Pneumonia; Lung Neoplasms; Pulmonary Embolism; Lung Diseases; Aortic Valve Stenosis

STUDY DESIGN:
Intervention Model Description: Randomization of patients referred for a CT scan of the thorax on one of three CT scanners routinely used for this purpose in our department
Masking Description: no masking required
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Scanner 1 (Other): Imaging performed on scanner 1: Photon-Counting Detector CT
  Interventions: Diagnostic Test: Imaging on Scanner with Spectral Imaging Capabilities
- Scanner 2 (Other): Imaging performed on scanner 2: Energy-Integrating Detector CT (128-slice)
  Interventions: Diagnostic Test: CT Scan using an Energy-Integrating Detector CT (128 slice MDCT)
- Scanner 3 (Other): Imaging performed on scanner 3: Energy-Integrating Detector CT (20-slice)
  Interventions: Diagnostic Test: CT Scan using an Energy-Integrating Detector CT (20-slice MDCT)

INTERVENTIONS:
Diagnostic Test: Imaging on Scanner with Spectral Imaging Capabilities — Patients will undergo imaging on a modern CT scanner with spectral imaging capabilities. A dose neutral spectral acquisition mode will routinely be used. Contrast material protocol and scan ranges are similar in all three arms.
  Other Names: CT Scan using a Photon-Counting Detector CT: Naeotom Alpha (Siemens Healthineers)
  Arms: Scanner 1
Diagnostic Test: CT Scan using an Energy-Integrating Detector CT (128 slice MDCT) — Patients will undergo imaging on a modern 128-slice CT scanner (Siemens Healthineers) with energy-integrating detector and without spectral acquisition mode. Contrast material protocol and scan ranges are similar in all three arms.
  Arms: Scanner 2
Diagnostic Test: CT Scan using an Energy-Integrating Detector CT (20-slice MDCT) — Patients will undergo imaging on a modern 20-slice CT scanner (Siemens Healthineers) with energy-integrating detector and without spectral acquisition mode. Contrast material protocol and scan ranges are similar in all three arms.
  Arms: Scanner 3

SUMMARY:
CT scans of the chest / thorax are of great importance both in the initial diagnosis and in the follow-up of pulmonary or thoracic diseases. As an example, CT angiography of the pulmonary arteries (CTPA) is worldwide considered to be gold standard test in patients with a suspicion for pulmonary embolism.

The aim of this study is to measure and compare dose efficiency of modern CT scanners for unenhanced and contrast-enhanced scan protocols of the chest/thorax. Patients who are referred for a CT of the chest/thorax will be randomly assigned to one of the three CT scanners currently in use at our institution.

ELIGIBILITY:
Inclusion Criteria:

* patient is referred for an unenhanced CT OR contrast-enhanced CT of the chest/thorax confirmed by a board-certified radiologist ('justifying indication' according to German/European radiation protection law) AND
* patient is at least 18 years of age AND
* patient (is able to give informed consent and) has given informed consent.

Exclusion Criteria:

* high degree of medical urgency (i.e. patient cannot be consented for iv contrast according to routine procedures)
* known or suspected pregnancy, or lactating . contraindications for contrast agent (renal failure, allergy, hyperthyroidism)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 958 (Actual)
Dates: Start 2021-10-07 (Actual); Primary Completion 2023-05-31 (Actual); Study Completion 2023-05-31 (Actual)

PRIMARY OUTCOMES:
Parameters of Objective Image Quality | 1 year
  Measured as signal, image noise and modulation transfer function equivalent parameters
Parameters of Radiation Dose | 1 year
  measured as x-ray tube parameters such as dose length product (DLP)

SECONDARY OUTCOMES:
Subjective Image Quality Evaluation (entire cohort and for individual disease groups) | 1 year
  measured by blinded evaluation by radiologists

CONTACTS AND LOCATIONS:
Overall Officials: Florian Schwarz, MD, Principal Investigator — Universitaetsklinikum Augsburg
Locations (1):
- University Hospital Augsburg, Augsburg, Bavaria, Germany

IPD SHARING:
Plan to Share IPD: Yes
We plan to share individual participant data upon request (pending final approval by the data protection officer).
Supporting Information: Study Protocol, SAP
Time Frame: Requests for sharing individual participant data will be considered at the time of publication of the first manuscript containing result data.
Access Criteria: We plan to share data on request at this point in time.